CLINICAL TRIAL: NCT00506207
Title: A Phase I and Pharmacokinetic Study of S-1 Combined With Irinotecan and Oxaliplatin in Advanced Gastrointestinal Malignancy
Brief Title: A Phase I Study of S-1 Plus Irinotecan and Oxaliplatin in Advanced Gastrointestinal Malignancy
Acronym: TIROX
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-166
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Colorectal Neoplasm; Gastric Neoplasm; Secondary
Keywords: Gastrointestinal neoplasms; Combination chemotherapy; S-1; Irinotecan; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis; Gastrointestinal Neoplasms | interventions — S 1 (combination); Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S-1, Irinotecan, Oxaliplatin

SUMMARY:
This study is an open-label, single center, and a dose-escalating phase I study to determine the maximal tolerated dose and the recommended dose of S-1 combined with irinotecan/oxaliplatin in patients with unresectable or metastatic colorectal or gastric carcinoma.

DETAILED DESCRIPTION:
Dose level and escalating schedule are followings;

* S-1 (level 1/2, 3/4, 5/6: 60, 70, 80 mg/m2/day) every 12-h p.o. on days 1(evening)-15 (morning)
* Irinotecan (level 1,2/3, 4/5, 6: 120, 130, 140, 150 mg/m2) mixed in d5w or normal saline 500 ml iv over 90 min on day 1
* Oxaliplatin 85 mg/m2 fixed dose mixed in d5w 250 ml iv infusion over 2-h on day 1

Treatment will be administered every 3 weeks. Start at dose level 1. Thereafter, dose level 2, 3, 4, 5, and 6. If dose-limiting toxicity (DLT) occurs at dose level 1, dose level at -1 will follow

Dose escalation will be continued until more than one-third of the patients in a given cohort show dose-limiting toxicity (DLT) during treatment cycle 1. At least three patients will be enrolled in each cohort. Before escalating to the next dose level, all three patients should have received at least one treatment cycle. If none of the first three treated patients develops DLT in the first cycle at a specific dose level, dose escalation will be continued. If one of the first three treated patients develops DLT at any dose level, then three additional patients are to be entered on the same dose level. If only one in six patients at a given level experiences a DLT, escalation will proceed. The MTD is defined as the dose level at which at least one-third of patients experienced a DLT. The RD for the subsequent phase II study is defined as the preceding dose level before the MTD is attained. Intra-patient dose escalation will not be permitted. Treatment will be continued in the absence of disease progression or unacceptable toxicity with maximum 12 cycles. For purpose of determining the MTD, only DLT occurring during the first cycle of therapy will be considered.

DLTs are defined as any of following;

* Grade 4 neutropenia lasting at least 7 days or grade 3 or 4 neutropenia associated with fever  38.3C as single axillary temperature or 38 C for 1-h
* Grade 4 thrombocytopenia
* Grade 3 or 4 non-hematological toxicity except alopecia, and nausea/vomiting
* Grade 3 or 4 nausea/vomiting not reduced to grade 1 with aggressive antiemetic support
* Inability of the patient to take 75% of the planned chemotherapy dose during the treatment period

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable or metastatic colorectal or gastric carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease, according to the RECIST criteria or non-measurable disease Measurable lesions
* Previous adjuvant, palliative chemotherapy including 5-FU, oxaliplatin and irinotecan, molecular targeted therapy and/or radiotherapy is allowed
* Adequate major organ functions
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Prior history of peripheral neuropathy
* Inadequate cardiovascular
* Serious concurrent infection or nonmalignant illness
* Other malignancy within the past 3 years except non-melanomatous skin cancer or carcinoma in situ of the cervix
* Psychiatric disorder that would preclude compliance
* Pregnant, nursing women or patients with reproductive potential without contraception
* Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or warfarin et al.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity measured by NCICTC v.3 | During treatment
Blood level of irinotecan and S-1 and their metabolites | At 1st cycle

SECONDARY OUTCOMES:
Maximal response rate, progression-free survival, survival

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, M.D.Ph.D, Principal Investigator
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea